CLINICAL TRIAL: NCT05712954
Title: The Effect of Using Music and Natural Landscape Paintings on Women's Pain Level, Anxiety and Analgesic Use During Hysterosalpingography
Brief Title: The Effect of Using Music and Natural Landscape Paintings on Pain Level, Anxiety and Analgesic Use of Women During HSG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ŞERİVAN KARAKUT (Other)
Responsible Party: Sponsor-Investigator, ŞERİVAN KARAKUT, lecturer, Hasan Kalyoncu University
Organization: Hasan Kalyoncu University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2022/126
Record Dates: First submitted 2022-12-30; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Hysterosalpingography; Anxiety; Pain
Keywords: hsg; music; natural landscape; anxiety
MeSH Terms: conditions — Anxiety Disorders; Pain; Charcot-Marie-Tooth Disease, Axonal, Type 2A2

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial model with pretest-posttest control group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (No Intervention): The study will start with the women in the control group. The women in the control group, who were selected in accordance with the sample selection criteria and agreed to be a participant, will be given data collection tools for the pre-test on the day of the procedure and no intervention will be made other than the counseling given at the hospital. VAS and State-Trait Anxiety Inventory will be applied after the procedure. After 24 hours, the women will be reached and questioned whether they use analgesics.
- music group (Experimental): The women in the 1st group will be pre-tested with data collection tools before the HSG, then after they are taken to the table, headphones will be put on and music will be played. VAS and State-Trait Anxiety Inventory will be applied after the procedure. After 24 hours, the women will be reached and questioned whether they use analgesics. After the women in this group are completed, the 2nd group will be started.
  Interventions: Other: music group
- video group (Experimental): 2. The women in the group will be pre-tested with data collection tools before the HSG, and after they are taken to the table, a video with natural landscape pictures prepared by the researcher will be opened on the iPad. VAS and State-Trait Anxiety Inventory will be applied after the procedure. After 24 hours, the women will be reached and questioned whether they use analgesics.
  Interventions: Other: video group

INTERVENTIONS:
Other: music group — music
  Arms: music group
Other: video group — video
  Arms: video group

SUMMARY:
The study was planned as a randomized controlled study in order to evaluate the use of music and natural scenery paintings in women who underwent HSG procedure, their pain level, anxiety and post-procedure analgesic use.

DETAILED DESCRIPTION:
The universe of the research; Women who apply to Dicle University Hospital's Obstetrics and Gynecology Polyclinic will be recommended to have an HSG.

Sample of the research:

Women who applied to the Dicle University Hospital Obstetrics and Gynecology Outpatient Clinic and recommended to have an HSG will participate in the study.

In the calculation of the sample size of the research, in the calculation made in line with the data taken from the reference studies; The sample size was used at the 95% confidence interval, the effect size was 0.80, and the alpha was 0.05, and it was seen that at least 29 individuals should be included in each group.

Application of Research The study was planned to be conducted on women who were recommended to have an HSG, who applied to the Dicle University Hospital Obstetrics and Gynecology Clinic between January 2022 and July 2023 in a randomized controlled manner. The Socio-Demographic Data Questionnaire, Visual Pain Scale, State-Trait Anxiety Inventory, and the Socio-Demographic Data Questionnaire, prepared by the researcher for the women who were selected in accordance with the sample selection criteria and accepted to be a participant, in line with the recommendations of the academicians specialized in the field of Gynecology and Gynecology Nursing. Analgesia Follow-up Form will be applied.

After the control group study is completed, the case group study will begin. The reason why the control and case groups were not studied at the same time was because it was thought that women saw each other and would be affected by each other.

In the control group, only the pre-test before the procedure, the post-test after the procedure and the use of analgesics within 24 hours after the HSG will be questioned with data collection tools and no attempt will be made.

Case groups will be pre-tested before the procedure, they will be listened to music or shown pictures of natural landscapes during the procedure, and after the procedure is completed, the post-test will be applied and 24 hours after the procedure, they will be contacted and questioned whether they use analgesics.

ELIGIBILITY:
Inclusion Criteria:

* In the research be over 18 years old
* At least primary school graduate
* Not have a diagnosed psychiatric illness
* Not having mental deficiency and communication problems
* No drug sensitivity or allergy
* Not having received infertility treatment before
* Being diagnosed with primary infertility

Exclusion Criteria:

* To be illiterate be under the age of 18
* Having a diagnosed psychiatric illness
* Mental disability and communication problems
* Having drug sensitivity and allergy
* Being diagnosed with secondary infertility

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2023-01-13 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Listening to Music During HSG Affects Women's Pain Level. | Up to 7 Months
  A visual analog scale will be applied to measure patients' pain. A state-continuity scale will be applied to measure their anxiety.Visual Analog Scale (VAS) It was developed to determine the pain levels of sick individuals . It is stated as a reproducible, sensitive and reliable method for assessing pain severity. The individual marks a number from 0 to 10 on a 10-centimeter (cm) vertical or horizontal line. Zero (0) means no pain, and 10 means unbearable pain.State-Trait Anxiety Inventory The items of the scale are arranged in a four-point Likert type and thus the total score is obtained. There are also negative and positive statements in the scale. In order to obtain the total scale score, the sum of the negative items is subtracted from the total of the positive items. The total score of the scale varies between 20 and 80, and a high score means that the individual has a high level of anxiety.

SECONDARY OUTCOMES:
Listening to Music During HSG Affects Women's Anxiety. | Up to 7 Months
  A visual analog scale will be applied to measure patients' pain. A state-continuity scale will be applied to measure their anxiety.Visual Analog Scale (VAS) It was developed to determine the pain levels of sick individuals . It is stated as a reproducible, sensitive and reliable method for assessing pain severity. The individual marks a number from 0 to 10 on a 10-centimeter (cm) vertical or horizontal line. Zero (0) means no pain, and 10 means unbearable pain.State-Trait Anxiety Inventory The items of the scale are arranged in a four-point Likert type and thus the total score is obtained. There are also negative and positive statements in the scale. In order to obtain the total scale score, the sum of the negative items is subtracted from the total of the positive items. The total score of the scale varies between 20 and 80, and a high score means that the individual has a high level of anxiety.

OTHER OUTCOMES:
Listening to Music During HSG Effective on Women's Analgesic Use. | Up to 7 Months
  A visual analog scale will be applied to measure patients' pain. A state-continuity scale will be applied to measure their anxiety.Visual Analog Scale (VAS) It was developed to determine the pain levels of sick individuals . It is stated as a reproducible, sensitive and reliable method for assessing pain severity. The individual marks a number from 0 to 10 on a 10-centimeter (cm) vertical or horizontal line. Zero (0) means no pain, and 10 means unbearable pain.State-Trait Anxiety Inventory The items of the scale are arranged in a four-point Likert type and thus the total score is obtained. There are also negative and positive statements in the scale. In order to obtain the total scale score, the sum of the negative items is subtracted from the total of the positive items. The total score of the scale varies between 20 and 80, and a high score means that the individual has a high level of anxiety.
Natural Landscape Pictures are Effective on the Pain Level of Women during HSG. | Up to 7 Months
  A visual analog scale will be applied to measure patients' pain. A state-continuity scale will be applied to measure their anxiety.Visual Analog Scale (VAS) It was developed to determine the pain levels of sick individuals . It is stated as a reproducible, sensitive and reliable method for assessing pain severity. The individual marks a number from 0 to 10 on a 10-centimeter (cm) vertical or horizontal line. Zero (0) means no pain, and 10 means unbearable pain.State-Trait Anxiety Inventory The items of the scale are arranged in a four-point Likert type and thus the total score is obtained. There are also negative and positive statements in the scale. In order to obtain the total scale score, the sum of the negative items is subtracted from the total of the positive items. The total score of the scale varies between 20 and 80, and a high score means that the individual has a high level of anxiety.
Natural Landscape Paintings Are Effective On Anxiety Level Of Women During HSG. | Up to 7 Months
  A visual analog scale will be applied to measure patients' pain. A state-continuity scale will be applied to measure their anxiety.Visual Analog Scale (VAS) It was developed to determine the pain levels of sick individuals . It is stated as a reproducible, sensitive and reliable method for assessing pain severity. The individual marks a number from 0 to 10 on a 10-centimeter (cm) vertical or horizontal line. Zero (0) means no pain, and 10 means unbearable pain.State-Trait Anxiety Inventory The items of the scale are arranged in a four-point Likert type and thus the total score is obtained. There are also negative and positive statements in the scale. In order to obtain the total scale score, the sum of the negative items is subtracted from the total of the positive items. The total score of the scale varies between 20 and 80, and a high score means that the individual has a high level of anxiety.
Natural Landscape Paintings During HSG Are Effective in Women's Use of Analgesics. | Up to 7 Months
  A visual analog scale will be applied to measure patients' pain. A state-continuity scale will be applied to measure their anxiety.Visual Analog Scale (VAS) It was developed to determine the pain levels of sick individuals . It is stated as a reproducible, sensitive and reliable method for assessing pain severity. The individual marks a number from 0 to 10 on a 10-centimeter (cm) vertical or horizontal line. Zero (0) means no pain, and 10 means unbearable pain.State-Trait Anxiety Inventory The items of the scale are arranged in a four-point Likert type and thus the total score is obtained. There are also negative and positive statements in the scale. In order to obtain the total scale score, the sum of the negative items is subtracted from the total of the positive items. The total score of the scale varies between 20 and 80, and a high score means that the individual has a high level of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Şerivan, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No